CLINICAL TRIAL: NCT05936294
Title: Cardiac Resynchronization Therapy With Synchronized RV Pacing to Improve Cardiac Function in Patients With Right Bundle Branch Block and Systolic LV Dysfunction
Brief Title: Adaptive Cardiac Resynchronization Therapy in Patients With RBBB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Henry Ford Health System (Other)
Collaborators: Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Waddah Maskoun, MD. Senior Staff Physician, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E17154
Record Dates: First submitted 2019-08-07; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Right Bundle-Branch Block
MeSH Terms: conditions — Bundle-Branch Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CRT Optimization (Other): Each patient will have atrial pacing 10% higher than the sinus rate or atrial pacing at a rate of 60 bpm if significant sinus bradycardia is present. Each patient will have six ECGs and echocardiographic sequences performed in the same session. In addition six electrical activation evaluations by the Medtronic ECG belt will be done as well. The first study will always be with no ventricular pacing. One study will be echocardiography-optimized BIV pacing and four studies for echocardiography-optimized (?) adaptive RV-only pacing with different AV intervals. A random-sequence will be performed to determine the order for the rest of the studies.
  Interventions: Diagnostic Test: Optimization of CRT Device

INTERVENTIONS:
Diagnostic Test: Optimization of CRT Device — Each patient will have atrial pacing 10% higher than the sinus rate or atrial pacing at a rate of 60 bpm if significant sinus bradycardia is present. Each patient will have six ECGs and echocardiographic sequences performed in the same session. In addition six electrical activation evaluations by the Medtronic ECG belt will be done as well. The first study will always be with no ventricular pacing. One study will be echocardiography-optimized BIV pacing and four studies for echocardiography-optimized (?) adaptive RV-only pacing with different AV intervals. A random-sequence will be performed to determine the order for the rest of the studies.

SUMMARY:
This study will address whether acute adaptive RV pacing in sinus rhythm patients with severe LV systolic dysfunction and RBBB is superior to no ventricular pacing, and is as effective as echocardiographically optimized biventricular (BIV) pacing based on Medtronic ECG belt and cardiac performance as assessed by the echocardiographic parameters of RV and LV function.

DETAILED DESCRIPTION:
Current guidelines state that CRT implantation is less beneficial for patients with RBBB compared to those with LBBB (2). Current evidence suggests that frequent or persistent RV-only pacing in patients with narrow QRS and LV dysfunction can be harmful due to ventricular desynchronization attributable to RV apex pacing (3-5).

Studies suggest that LV-only pacing is not inferior to BIV pacing in sinus rhythm patients with LV dysfunction and LBBB and ICD back up (6,7). A novel algorithm of CRT by delivering synchronized LV pacing with the intrinsic conduction in patients with severe LV systolic dysfunction and LBBB (adaptive CRT) has been demonstrated to show that it is at least as effective as protocol-driven echocardiographic optimization. It also has shown a significant reduction in the probability of 30-day readmission for both HF and all-cause hospitalizations, 46% reduced incidence of AF compared to conventional CRT, and prolongation of CRT device battery life (8-10). Patients who had an adaptive CRT algorithm that provided > 50% synchronized LV pacing or had normal AV conduction with the adaptive CRT algorithm had decreased risk of death or heart failure hospitalization when compared to those with <50% synchronized LV pacing or echocardiography-optimized BIV pacing respectively (11). In another acute study the LV dP/dtmax was higher with LV than BIV pacing when LV pacing was associated with ventricular fusion caused by intrinsic activation (12).

Several studies have suggested that optimization of the programmed atrioventricular delay (AVD) and interventricular delay (VVD) delays may incrementally improve the long-term outcome of BIV pacing (13-15).

The lateral LV wall contracts early in patients with RBBB when compared to LBBB so LV pacing in the CRT devices is less likely to be beneficial. . In an experimental study of 12 dogs with tachycardia-induced cardiomyopathy and RBBB (6 dogs) or LBBB (6 dogs) (16), RV-only pacing enhanced LV function and synchrony as seen by dP/dtmax measured by catheter tip placed in the LV chamber and synchrony evaluation by cardiac MRI in the RBBB group as well or better than BIV pacing. LV-only pacing worsened function in the RBBB group.

RV-only pacing was also evaluated in a prospective study of 7 patients with RBBB and RV dysfunction with most patients having congenital heart disease. LV global function was intact at baseline (17). Sequential atrioventricular RV pacing with an atrioventricular delay of 90% of the PR interval was superior to atrial-only pacing for both improvement in RV dP/dtmax and LV cardiac index as seen at cardiac catheterization. The RV dP/dtmax increased by 22% in RBBB patients with RV pacing and QRS decreased from 163 +/- 39 to 126 +/- 31 ms. The two studies together suggest that most of the benefit from BIV pacing in patients with RBBB and HF is due to the RV pacing component and the benefit might be reduced due to the LV pacing component. Better timing of RV pacing in patients with RBBB might significantly decrease desynchronization from RV pacing and maximize the benefit of RV pacing as seen in adaptive LV-pacing CRT in patients with LBBB and LV systolic dysfunction.

These studies have led to the current hypothesis that adaptive RV pacing using RV-only pacing synchronized to LV activation when intrinsic AV conduction is normal is more physiological and will improve RV and LV function by Echocardiography parameters and on Medtronic ECG belt for activation in patients with RBBB and LV dysfunction because of improved synchronization and narrowing the QRS duration.

As a secondary goal, battery life with BIV pacing will be compared to adaptive RV pacing assuming at least 50% of RV-only pacing will be achieved with adaptive CRT for RBBB.

ELIGIBILITY:
Inclusion Criteria: Included patients will have:

* sinus rhythm or isolated atrial pacing
* LV systolic dysfunction (EF <35% at time of device implant)
* AV conduction <250 ms, RBBB, and
* have an implanted CRT device based on the ACC/AHA/HRS guidelines (2, 18) or will have a CRT device implanted during the study enrollment per ACC/AHA/HRS guidelines (2).

Exclusion Criteria:

* atrial fibrillation
* atrial flutter
* atrial tachycardia
* AV delay > 250 ms
* sinus tachycardia with resting heart rate at time of the study 100 bpm
* frequent APCs (> 25% of the total beats/min) or PVCs (>20% of the total beats/min), or
* patients with EF > 40% at time of enrollment (if LV systolic function was found to be improved from time of implant).

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of adaptive Right Ventricular (RV) pacing | 1 hour
  Echocardiographic parameters to measure cardiac function, including:
  1. Left Ventricular Outflow Tract velocity time interval(LVOT VTI),
  2. dP/dt of Left Ventricle (LV) and RV,
  3. Myocardial Performance Index (MPI),
  4. Right Ventricular Outflow Tractvelocity time interval (RVOT VTI); and
  5. 3D derived Systolic Dyssynchrony Index (SDI).

SECONDARY OUTCOMES:
Battery/device longevity | 1 hour
  Calculations of current drain and pacing percentages for RV-only pacing versus BIV pacing. Measured by microjoule current consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Waddah Maskoun, MD, Principal Investigator — Henry Ford
Locations (2):
- United States (2):
  - Central Arkansas Veterans Healthare System, Little Rock, Arkansas
  - Henry Ford Hospital, Detroit, Michigan

REFERENCES:
- [Background] Surawicz B, Childers R, Deal BJ, Gettes LS, Bailey JJ, Gorgels A, Hancock EW, Josephson M, Kligfield P, Kors JA, Macfarlane P, Mason JW, Mirvis DM, Okin P, Pahlm O, Rautaharju PM, van Herpen G, Wagner GS, Wellens H; American Heart Association Electrocardiography and Arrhythmias Committee, Council on Clinical Cardiology; American College of Cardiology Foundation; Heart Rhythm Society. AHA/ACCF/HRS recommendations for the standardization and interpretation of the electrocardiogram: part III: intraventricular conduction disturbances: a scientific statement from the American Heart Association Electrocardiography and Arrhythmias Committee, Council on Clinical Cardiology; the American College of Cardiology Foundation; and the Heart Rhythm Society. Endorsed by the International Society for Computerized Electrocardiology. J Am Coll Cardiol. 2009 Mar 17;53(11):976-81. doi: 10.1016/j.jacc.2008.12.013. No abstract available. PMID 19281930
- [Background] Tracy CM, Epstein AE, Darbar D, Dimarco JP, Dunbar SB, Estes NA 3rd, Ferguson TB Jr, Hammill SC, Karasik PE, Link MS, Marine JE, Schoenfeld MH, Shanker AJ, Silka MJ, Stevenson LW, Stevenson WG, Varosy PD. 2012 ACCF/AHA/HRS focused update of the 2008 guidelines for device-based therapy of cardiac rhythm abnormalities: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2012 Oct 2;60(14):1297-313. doi: 10.1016/j.jacc.2012.07.009. Epub 2012 Sep 10. No abstract available. PMID 22975230
- [Background] Wilkoff BL, Cook JR, Epstein AE, Greene HL, Hallstrom AP, Hsia H, Kutalek SP, Sharma A; Dual Chamber and VVI Implantable Defibrillator Trial Investigators. Dual-chamber pacing or ventricular backup pacing in patients with an implantable defibrillator: the Dual Chamber and VVI Implantable Defibrillator (DAVID) Trial. JAMA. 2002 Dec 25;288(24):3115-23. doi: 10.1001/jama.288.24.3115. PMID 12495391
- [Background] Steinberg JS, Fischer A, Wang P, Schuger C, Daubert J, McNitt S, Andrews M, Brown M, Hall WJ, Zareba W, Moss AJ; MADIT II Investigators. The clinical implications of cumulative right ventricular pacing in the multicenter automatic defibrillator trial II. J Cardiovasc Electrophysiol. 2005 Apr;16(4):359-65. doi: 10.1046/j.1540-8167.2005.50038.x. PMID 15828875
- [Background] Sharma AD, Rizo-Patron C, Hallstrom AP, O'Neill GP, Rothbart S, Martins JB, Roelke M, Steinberg JS, Greene HL; DAVID Investigators. Percent right ventricular pacing predicts outcomes in the DAVID trial. Heart Rhythm. 2005 Aug;2(8):830-4. doi: 10.1016/j.hrthm.2005.05.015. PMID 16051118
- [Background] Boriani G, Gardini B, Diemberger I, Bacchi Reggiani ML, Biffi M, Martignani C, Ziacchi M, Valzania C, Gasparini M, Padeletti L, Branzi A. Meta-analysis of randomized controlled trials evaluating left ventricular vs. biventricular pacing in heart failure: effect on all-cause mortality and hospitalizations. Eur J Heart Fail. 2012 Jun;14(6):652-60. doi: 10.1093/eurjhf/hfs040. Epub 2012 Apr 17. PMID 22510423
- [Background] Boriani G, Kranig W, Donal E, Calo L, Casella M, Delarche N, Lozano IF, Ansalone G, Biffi M, Boulogne E, Leclercq C; B-LEFT HF study group. A randomized double-blind comparison of biventricular versus left ventricular stimulation for cardiac resynchronization therapy: the Biventricular versus Left Univentricular Pacing with ICD Back-up in Heart Failure Patients (B-LEFT HF) trial. Am Heart J. 2010 Jun;159(6):1052-1058.e1. doi: 10.1016/j.ahj.2010.03.008. PMID 20569719
- [Background] Martin DO, Lemke B, Birnie D, Krum H, Lee KL, Aonuma K, Gasparini M, Starling RC, Milasinovic G, Rogers T, Sambelashvili A, Gorcsan J 3rd, Houmsse M; Adaptive CRT Study Investigators. Investigation of a novel algorithm for synchronized left-ventricular pacing and ambulatory optimization of cardiac resynchronization therapy: results of the adaptive CRT trial. Heart Rhythm. 2012 Nov;9(11):1807-14. doi: 10.1016/j.hrthm.2012.07.009. Epub 2012 Jul 14. PMID 22796472
- [Background] Gasparini M, Birnie D, Lemke B, Aonuma K, Lee KL, Gorcsan J 3rd, Landolina M, Klepfer R, Meloni S, Cicconelli M, Grammatico A, Martin DO. Adaptive Cardiac Resynchronization Therapy Reduces Atrial Fibrillation Incidence in Heart Failure Patients With Prolonged AV Conduction: The Adaptive CRT Randomized Trial. Circ Arrhythm Electrophysiol. 2019 May;12(5):e007260. doi: 10.1161/CIRCEP.119.007260. No abstract available. PMID 30991823
- [Background] Starling RC, Krum H, Bril S, Tsintzos SI, Rogers T, Hudnall JH, Martin DO. Impact of a Novel Adaptive Optimization Algorithm on 30-Day Readmissions: Evidence From the Adaptive CRT Trial. JACC Heart Fail. 2015 Jul;3(7):565-572. doi: 10.1016/j.jchf.2015.03.001. Epub 2015 Jun 10. PMID 26071616
- [Background] Birnie D, Lemke B, Aonuma K, Krum H, Lee KL, Gasparini M, Starling RC, Milasinovic G, Gorcsan J 3rd, Houmsse M, Abeyratne A, Sambelashvili A, Martin DO. Clinical outcomes with synchronized left ventricular pacing: analysis of the adaptive CRT trial. Heart Rhythm. 2013 Sep;10(9):1368-74. doi: 10.1016/j.hrthm.2013.07.007. Epub 2013 Jul 11. PMID 23851059
- [Background] van Gelder BM, Bracke FA, Meijer A, Pijls NH. The hemodynamic effect of intrinsic conduction during left ventricular pacing as compared to biventricular pacing. J Am Coll Cardiol. 2005 Dec 20;46(12):2305-10. doi: 10.1016/j.jacc.2005.02.098. PMID 16360063
- [Background] Sawhney NS, Waggoner AD, Garhwal S, Chawla MK, Osborn J, Faddis MN. Randomized prospective trial of atrioventricular delay programming for cardiac resynchronization therapy. Heart Rhythm. 2004 Nov;1(5):562-7. doi: 10.1016/j.hrthm.2004.07.006. PMID 15851220
- [Background] Morales MA, Startari U, Panchetti L, Rossi A, Piacenti M. Atrioventricular delay optimization by doppler-derived left ventricular dP/dt improves 6-month outcome of resynchronized patients. Pacing Clin Electrophysiol. 2006 Jun;29(6):564-8. doi: 10.1111/j.1540-8159.2006.00402.x. PMID 16784420
- [Background] Vidal B, Sitges M, Marigliano A, Delgado V, Diaz-Infante E, Azqueta M, Tamborero D, Tolosana JM, Berruezo A, Perez-Villa F, Pare C, Mont L, Brugada J. Optimizing the programation of cardiac resynchronization therapy devices in patients with heart failure and left bundle branch block. Am J Cardiol. 2007 Sep 15;100(6):1002-6. doi: 10.1016/j.amjcard.2007.04.046. Epub 2007 Jul 5. PMID 17826387
- [Background] Byrne MJ, Helm RH, Daya S, Osman NF, Halperin HR, Berger RD, Kass DA, Lardo AC. Diminished left ventricular dyssynchrony and impact of resynchronization in failing hearts with right versus left bundle branch block. J Am Coll Cardiol. 2007 Oct 9;50(15):1484-90. doi: 10.1016/j.jacc.2007.07.011. Epub 2007 Sep 24. PMID 17919569
- [Background] Dubin AM, Feinstein JA, Reddy VM, Hanley FL, Van Hare GF, Rosenthal DN. Electrical resynchronization: a novel therapy for the failing right ventricle. Circulation. 2003 May 13;107(18):2287-9. doi: 10.1161/01.CIR.0000070930.33499.9F. Epub 2003 May 5. PMID 12732607
- [Background] Epstein AE, DiMarco JP, Ellenbogen KA, Estes NA 3rd, Freedman RA, Gettes LS, Gillinov AM, Gregoratos G, Hammill SC, Hayes DL, Hlatky MA, Newby LK, Page RL, Schoenfeld MH, Silka MJ, Stevenson LW, Sweeney MO, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Buller CE, Creager MA, Ettinger SM, Faxon DP, Halperin JL, Hiratzka LF, Hunt SA, Krumholz HM, Kushner FG, Lytle BW, Nishimura RA, Ornato JP, Page RL, Riegel B, Tarkington LG, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the ACC/AHA/NASPE 2002 Guideline Update for Implantation of Cardiac Pacemakers and Antiarrhythmia Devices); American Association for Thoracic Surgery; Society of Thoracic Surgeons. ACC/AHA/HRS 2008 Guidelines for Device-Based Therapy of Cardiac Rhythm Abnormalities: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the ACC/AHA/NASPE 2002 Guideline Update for Implantation of Cardiac Pacemakers and Antiarrhythmia Devices): developed in collaboration with the American Association for Thoracic Surgery and Society of Thoracic Surgeons. Circulation. 2008 May 27;117(21):e350-408. doi: 10.1161/CIRCUALTIONAHA.108.189742. Epub 2008 May 15. No abstract available. PMID 18483207
- [Background] Krum H, Lemke B, Birnie D, Lee KL, Aonuma K, Starling RC, Gasparini M, Gorcsan J, Rogers T, Sambelashvili A, Kalmes A, Martin D. A novel algorithm for individualized cardiac resynchronization therapy: rationale and design of the adaptive cardiac resynchronization therapy trial. Am Heart J. 2012 May;163(5):747-752.e1. doi: 10.1016/j.ahj.2012.02.007. PMID 22607850
- [Background] Lane RE, Chow AW, Chin D, Mayet J. Selection and optimisation of biventricular pacing: the role of echocardiography. Heart. 2004 Dec;90 Suppl 6(Suppl 6):vi10-6. doi: 10.1136/hrt.2004.043000. PMID 15564419
- [Background] Ypenburg C, Van De Veire N, Westenberg JJ, Bleeker GB, Marsan NA, Henneman MM, Van Der Wall EE, Schalij MJ, Abraham TP, Barold SS, Bax JJ. Noninvasive imaging in cardiac resynchronization therapy--Part 2: Follow-up and optimization of settings. Pacing Clin Electrophysiol. 2008 Dec;31(12):1628-39. doi: 10.1111/j.1540-8159.2008.01237.x. PMID 19067818